CLINICAL TRIAL: NCT03684005
Title: MyPatientPal: An App to Help Patients Manage Their Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Felicity Harper (Other)
Responsible Party: Sponsor-Investigator, Felicity Harper, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-063
Record Dates: First submitted 2018-09-22; First posted 2018-09-25 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Smartphone App Use (Other): All patients in this single-arm study will use a smartphone-based app, MyPatientPal, to enter symptoms and track medications related to their cancer treatment. No drugs will be administered for the purposes of this behavioral study.
  Interventions: Other: MyPatientPal smartphone app

INTERVENTIONS:
Other: MyPatientPal smartphone app — All patients in this single-arm study will use a smartphone-based app, MyPatientPal, to enter symptoms and track medications related to their cancer treatment. No drugs will be administered for the purposes of this behavioral study.

SUMMARY:
MyPatientPal was developed in collaboration with both patient and oncologist stakeholders, is designed to facilitate such patient self-management through the daily reporting of side effects and medications.

DETAILED DESCRIPTION:
MyPatientPal is a patient app that is designed to help patients track and manage treatment side effects and medication adherence on a daily basis. Side effects (e.g., pain, fatigue, diarrhea, nausea) can be physically and emotionally debilitating, and when uncontrolled, can cause treatment complications, resulting in unscheduled care costs, patient out-of-pocket costs, and delays or discontinuation of treatment. The app allows personalization of daily entries such that patients can select the specific medications and dosage and side effects (using items from the NCI Common Terminology Criteria for Adverse Events) that they and/or their providers want to track. A charting feature provides an easy-to-read display of patients' daily reports, summarizing the intensity and frequency of side effects and medication use either by week or by month. These reports can also be printed out and shared with providers.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of any solid tumor cancer
* Be starting treatment using an oral cancer therapeutic agent
* Be able to speak, read, and write English
* Willing and able to use their smartphone to use MyPatientPal

Exclusion Criteria:

* Patients with cognitive or perceptual disturbances

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Treatment-related symptoms | Symptoms will be reported weekly via the internet for weeks 1-4 and daily for weeks 5-8 via the smartphone app
  The frequency of treatment-related symptoms will be examined as the primary outcome. Patients will report the frequency and severity of symptoms selected from a symptom survey that consists of a list of 17 symptoms derived from the National Cancer Institute (NCI) CTCAE (Common Terminology Criteria for Adverse Events). Examples include diarrhea, constipation, vomiting, fever, and fatigue. Patients will be asked to mark the frequency of each symptom using a 5-point rating scale (from 0=none to 4=very severe). A total symptom impact score will be calculated by summing item responses across all symptoms. The investigators will compare the overall mean difference between the weekly and daily reporting phases.

SECONDARY OUTCOMES:
Adherence to medications | Adherence will be reported weekly via the internet for weeks 1-4 and daily for weeks 5-8 via the smartphone app
  Patient adherence to oral chemotherapy will be examined as a secondary outcome. Patients will report any medications they are taking related to their treatment. Each report will consist of them answering a forced-choice question about whether each of their self-selected medications was taken (0=yes, 1=no). The investigators will compare the ratio of total days of adherence/total number of days per medication between the weekly and daily reporting phases. There will be no set number of medications that will be assessed given that patients will self-select their own medications, but on average, patients will report on 3 medications. Examples may include Xeloda, Ibrance, Femara, Tamoxifen, Remeron, Reglan, or Compazine.
Patient self-efficacy | Patient self-efficacy will be reported weekly via the internet for weeks 1-4 and daily for weeks 5-8 via the smartphone app
  Patient self-efficacy will be examined as a secondary outcome. Patient self-efficacy for managing treatment side effects will be assessed with a 13-item version of the Chronic Pain Self-Efficacy Scale, which has been modified for a cancer population. Items assess patients' self-efficacy for managing and coping with side effects. Examples are "How certain is the participant that they can control their fatigue?" and "How certain is the participant that they can cope with mild to moderate pain?" Items are rated on a 10-point Likert scale ranging from 10 = very uncertain and 100 = very certain and items scores are summed for a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Felicity Harper, PhD, Principal Investigator — Associate Professor/PI
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No